CLINICAL TRIAL: NCT06642883
Title: Evaluation of the Effects of 10-strain Probiotic (ProLife 10 FORTE) on Gut Microbiota Composition in Patients Presenting with Ulcerative Colitis During the Remission Phase
Brief Title: Evaluation of ProLife 10 FORTE on Gut Microbiota Composition in UC Patients
Acronym: ProZ-UC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Savarino Edoardo Vincenzo, Prof, University of Padova
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5890/AO/23
Record Dates: First submitted 2024-09-09; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Ulcerative Colitis in Remission
Keywords: Microbiota, Probiotics

STUDY DESIGN:
Intervention Model Description: This is a double-blind, placebo-controlled, randomized trial in which the enrolled subjects will be included in one year. After the written informed consent collection, subjects will be randomized in a 1:1 ratio to the Group 1 or Group 2:
  * Group 1 will take Treatment A: 1 vial/day of PROLIFE 10 FORTE for 60 days.
  * Group 2 will take the Treatment B: 1 vial/day of placebo for 60 days.
  We will enroll 70 UC patients in the remission phase, both males and females, with a diagnosis of Ulcerative Colitis for at least three months. The therapy undertaken could not be changed nor stopped during the probiotic administration
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prolife 10 Forte (Active Comparator): Treatment: 1 dose/die (contains 10 ml with: in particular, 7 strains of Lactobacillus (L. casei R215, L. plantarum Lp-115, L. helveticus R0052, L. acidophilus La-14, L. gasseri Lg-36, L. brevis Lbr-35, L. rhamnosus HN001), 2 strains of Bifidobacteria (B. lactis Bl-04 and HN019) and Bacillus coagulans BC4. In addition, it contains 10 mg of glucoligosaccharide and a pool of Vitamin B (B1, B2, B6, B12).
  Interventions: Dietary Supplement: Prolife
- Placebo (Placebo Comparator): Treatment 1dose/die ( All additional components except probiotics and vitamins)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Prolife — randomized in a 1:1 ratio to treatment :1 vial/day for 60 days.
  Arms: Prolife 10 Forte
Dietary Supplement: Placebo — Placebo: 1 vial/day for 60 days.
  Arms: Placebo

SUMMARY:
This clinical trial aims to learn if the probiotic Prolife 10 Forte could improve the Gut Microbiota composition of Ulcerative colitis patients during the remission phase. The main questions it seeks to answer are:

* Does Prolife 10 Forte improve the microbiota composition in patients with Ulcerative colitis?
* Is it possible to highlight the variation in microbial pathways?
* What clinical parameters vary and are associated with changes in the gut microbiota? Researchers will compare Prolife 10 Forte to a placebo (a look-alike substance containing no drug) to see if the probiotics improve microbiota.

Participants will:

* Take 1 vial/day of Prolife 10 Forte /Placebo for 60 days.
* Visit the clinic two times for checkups, Questionaire and tests

DETAILED DESCRIPTION:
Ulcerative colitis (UC) is a chronic, idiopathic inflammatory disease that affects the colon. It is characterized by relapsing and remitting mucosal inflammation, and it can either affect only the rectum or extend along the colon. It is known that the gut microbiota also affects UC pathology. When its composition is altered, some microbiota-dependent mechanisms may be lost, resulting in an unbalanced relationship with the host: this condition is known with the name dysbiosis.Differences in gut microbiome composition and function have been associated with a variety of chronic diseases ranging from gastrointestinal inflammatory and metabolic conditions to neurological, cardiovascular, and respiratory illnesses.

Some trials have already been performed to understand if probiotics can also help in the UC management. For what concerns the human population, the literature contains many studies performed to evaluate the effect of different products on active or remitting disease. Most of the available literature is related to the use of a multiple-strain probiotic demonstrated that probiotic strains led to remission in some UC patients, with significant improvement in rectal bleeding and stool frequency, mucosal appearance, and clinical evaluation.

Prolife 10 FORTE has already been tested by our team to evaluate its composition and its ability to reach the gut, with positive results (unpublished data). Our team has performed the Shotgun analysis of the Prolife 10 FORTE that has confirmed the presence of all 10 strains of probiotics. The metabolic parameters of the product were also analyzed, highlighting a potential enrichment in the production of SCFA and in the fermentative pathways' degradation of starches, the biosynthesis of deoxyribonucleotides, and vitamins B2, B9, K, etc...

Thus, considering these positive premises, we now want to verify if Prolife 10 FORTE could improve the Gut Microbiota composition of UC patients during the remission phase.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of UC confirmed by clinical, endoscopic, and histopathological evidence. Disease in remission phase confirmed by clinical, endoscopic, and histopathological evidence.
* Age between 18 and 75 years old.
* Ability of the subject to participate fully in all aspects of this clinical trial.

Exclusion Criteria:

* Patients with active UC are determined by clinical, endoscopic, and histopathological evidence.
* Known diagnosis of CD, indeterminate colitis, ischemic colitis, radiation colitis, diverticular disease associated with colitis or microscopic colitis.
* Positive stool culture for active C. difficile.
* Pregnant women.
* Allergy to soy or fructose (contained in Prolife 10 FORTE)
* Patients under antibiotic and/or probiotic treatment within 10 days before visit1.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the gut microbiota composition variation (microbiota test) | From enrollment to the end of treatment 8 weeks
  Collection of fecal samples to assess the fecal microbiota composition ( rRNA16S) The 16S rRNA gene is a bacterial ribosomal gene and a part of the 30S subunit used in the identification, characterization, and classification of various bacteria. Samples were normalized, pooled, and run on Illumina MiSeq, to evaluate the composition of gut microbiota in terms of bacterial diversity ( alfa and beta) and abundance and any variability associated with the treatment.

SECONDARY OUTCOMES:
Evaluation of gut microbiota pathways variation ( Picrust analysis) | The microbiota analysis period, after 16S analysis: 2 months
  PICRUSt (Phylogenetic Investigation of Communities by Reconstruction of Unobserved States) is a bioinformatics tool used to predict the genetic functions of microbial communities based on DNA sequencing data.

OTHER OUTCOMES:
Evaluation of clinical parameters variation ( Fecal calprotectin stool test) | From enrolment to the end of analysis: 2-3 months
  The patient undergoes fecal calprotectin analysis assessment before and after the 60-day treatment. (cut-off value 50ug/g)
Evaluation of clinical parameters (IBDQ-32 questionnaire) | from the enrolment to the end of analysis: 2-3 months
  The patient undergoes IBDQ questionnaire assessment before and after the 60-day treatment. ( IBDQ-32 score; cut-off 170 pt.)

CONTACTS AND LOCATIONS:
Overall Officials: Edoardo V Savarino, Principal Investigator — University of Padova
Locations (1):
- Edoardo Vincenzo Savarino, Padua, Padua, Italy

IPD SHARING:
Plan to Share IPD: No